CLINICAL TRIAL: NCT02704442
Title: Does Anxiety in Children on the Day of Surgery Impact Compliance in the Ophthalmology Clinic?
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Queen's University (Other)
Collaborators: University of Regina (Other)
Responsible Party: Principal Investigator, Dr. Rachel Rooney, Rachel Rooney MD FRCPC, Assistant Professor Department of Anesthesiology, Queen's University, Queen's University
Other Study IDs: 6014969
Record Dates: First submitted 2016-02-17; First posted 2016-03-10 (Estimated); Last update posted 2018-04-26 (Actual); Status verified 2018-04

CONDITIONS: Anxiety; Strabismus; Compliance
Keywords: anesthesiology; ophthalmology
MeSH Terms: conditions — Anxiety Disorders; Strabismus; Patient Compliance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
The hypothesis is that pediatric patients with increased levels of anxiety on the day of surgery, in particular at point of anesthetic induction, will demonstrate decreased compliance with assessment in ophthalmology clinic postoperatively.

DETAILED DESCRIPTION:
There are many studies demonstrating pediatric anxiety from a surgical experience leading to postoperative maladaptive behaviors such as nightmares, separation anxiety, eating problems, and increased fear of doctors. There is a significant amount of research looking at day of surgery anxiety and pain in children and possible modifiers. Very little work has explored the effect of maladaptive behaviors with follow up physician visits. Strabismus surgery is particularly important as children require early and regular follow up assessments after surgery for optimal outcome. These assessments are meticulous and require good patient cooperation in order to obtain useful information for the pediatric ophthalmologist.

The study hypothesis is that pediatric patients with increased levels of anxiety on the day of surgery, in particular at point of anesthetic induction, will demonstrate decreased compliance with assessment in ophthalmology clinic postoperatively. The investigators expect this decrease in compliance will be evident based on changes seen on the ophthalmology clinic compliance scores generated pre and postoperatively.

The proposed study will be a prospective cross sectional study. Investigators will be measuring compliance in the ophthalmology clinic pre and postoperative and relating any changes in compliance with anxiety levels on the day of surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age 3 - 10 years old
* ASA I - III
* Primary strabismus surgery one or both eyes

Exclusion Criteria:

* Preexisting anxiety disorder
* Preexisting chronic pain or chronic analgesia use
* Neurobehavioural pathology limiting our ability to assess the patient eg: Cerebral Palsy, Autism or Developmental Delay.
* Inability to adhere to study protocol
* Consult in Anesthesiology clinic prior to surgery

Ages: 3 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Study personnel with approach all pediatric patients who are American Society of Anesthesia (ASA) classification I to III, between the ages of 3 and 10 attending the ophthalmology clinic for primary strabismus repair
Sampling Method: Non-Probability Sample
Enrollment: 82 (Estimated)
Dates: Start 2016-02; Primary Completion 2019-09 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
Change in Compliance with Ophthalmology examination | 4 days and 6 weeks after surgery
  A five point observer-rated Ophthalmology Clinic Compliance Checklist (OCCC) will be completed at the clinic visit one week prior to surgery and then at the 4 day and 6 week postoperative visits. The checklist includes sitting the ophthalmic chair, cover test, vision testing, stereo acuity and cycloplegic refraction. Compliance will be rated on a scale of 0 (non compliant ) 1 (compliant with minor coaxing) 2 (compliant with heavy coaxing) 3 (easily compliant)

SECONDARY OUTCOMES:
child observer rated anxiety | Observations on day of surgery at time points 1. admission to hospital 2. day surgery waiting area 3. just prior to entering the operating room 4. anesthetic induction 5. recovery room and at 4 days and 6 weeks post operatively
  Child observer-rated anxiety on day of surgery will be measured using the modified Yale Preoperative Anxiety Scale at 5 time-points throughout day-surgery process as described above and at Ophthalmology Clinic after surgery (i.e., day 4 post-surgery and 6 weeks post-surgery)
parent anxiety | measured at 4 time points: 1. at the last clinic visit prior to surgery (approximately 7 days), on day of surgery 2. at admission to hospital and 3. in the recovery room after surgery and 4. 4 days after surgery at the post op clinic visit
  Levels of parental anxiety will be measured by completion of the State-Trait Anxiety Inventory-state version at 3 time-points stated.
child temperament | pre operative assessment
  Parents will also be asked to complete a measure of child temperament [i.e., Emotionality, Activity, Sociability, Impulsivity temperament scale prior to the day of surgery (i.e., at clinic one week prior to surgery) 11.

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Rooney, MD, Principal Investigator — Queen's University
Locations (1):
- Hotel Dieu Hospital, Kingston, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kain ZN, Caldwell-Andrews AA. Preoperative psychological preparation of the child for surgery: an update. Anesthesiol Clin North Am. 2005 Dec;23(4):597-614, vii. doi: 10.1016/j.atc.2005.07.003. PMID 16310653
- [Background] Kain ZN, Mayes LC, Caldwell-Andrews AA, Karas DE, McClain BC. Preoperative anxiety, postoperative pain, and behavioral recovery in young children undergoing surgery. Pediatrics. 2006 Aug;118(2):651-8. doi: 10.1542/peds.2005-2920. PMID 16882820
- [Background] Kain ZN, Wang SM, Mayes LC, Caramico LA, Hofstadter MB. Distress during the induction of anesthesia and postoperative behavioral outcomes. Anesth Analg. 1999 May;88(5):1042-7. doi: 10.1097/00000539-199905000-00013. PMID 10320165
- [Background] Varughese AM, Nick TG, Gunter J, Wang Y, Kurth CD. Factors predictive of poor behavioral compliance during inhaled induction in children. Anesth Analg. 2008 Aug;107(2):413-21. doi: 10.1213/ane.0b013e31817e616b. PMID 18633018
- [Background] Kain ZN, Mayes LC, Wang SM, Caramico LA, Hofstadter MB. Parental presence during induction of anesthesia versus sedative premedication: which intervention is more effective? Anesthesiology. 1998 Nov;89(5):1147-56; discussion 9A-10A. doi: 10.1097/00000542-199811000-00015. PMID 9822003
- [Background] Wollin SR, Plummer JL, Owen H, Hawkins RM, Materazzo F. Predictors of preoperative anxiety in children. Anaesth Intensive Care. 2003 Feb;31(1):69-74. doi: 10.1177/0310057X0303100114. PMID 12635399
- [Background] Wright KD, Stewart SH, Finley GA. When are parents helpful? A randomized clinical trial of the efficacy of parental presence for pediatric anesthesia. Can J Anaesth. 2010 Aug;57(8):751-8. doi: 10.1007/s12630-010-9333-1. Epub 2010 May 25. PMID 20499223
- [Background] Kim JE, Jo BY, Oh HM, Choi HS, Lee Y. High anxiety, young age and long waits increase the need for preoperative sedatives in children. J Int Med Res. 2012;40(4):1381-9. doi: 10.1177/147323001204000416. PMID 22971489
- [Background] Kain ZN, Mayes LC, Cicchetti DV, Bagnall AL, Finley JD, Hofstadter MB. The Yale Preoperative Anxiety Scale: how does it compare with a "gold standard"? Anesth Analg. 1997 Oct;85(4):783-8. doi: 10.1097/00000539-199710000-00012. PMID 9322455